CLINICAL TRIAL: NCT04199325
Title: Probiotics for Gout / Hyperuricemia: A Randomized, Double-blind, Intervention, Parallel Controlled, Multicenter Clinical Trial
Brief Title: Probiotics for Gout / Hyperuricemia: A Randomized, Intervention, Parallel Controlled, Multicenter Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Collaborators: Inner Mongolia University of Science and Technology (Other); Inner Mongolia Hulunboir hospital (Unknown); Inner Mongolia People's Hospital (Other); Inner Mongolia Ordos Central Hospital (Unknown); Inner Mongolia Baogang Hospital (Other); Inner Mongolia Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: qpfff@126.com
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Gout; Hyperuricemia
Keywords: gout; hyperuricemia; probiotics
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Dietary Supplement: Probiotics; Drug: uric-acid-lowering drug
- Control group (Placebo Comparator)
  Interventions: Drug: uric-acid-lowering drug

INTERVENTIONS:
Dietary Supplement: Probiotics — Patients will be randomly assigned to the routine treatment + placebo group and probiotics + routine treatment group according to 1:2 ratio.
  Arms: Intervention group
Drug: uric-acid-lowering drug — Patients will be randomly assigned to the routine treatment + placebo group and probiotics + routine treatment group according to 1:2 ratio.

SUMMARY:
Under the premise of double-blind and non-interference clinical treatment, to evaluate the clinical efficacy and safety of probiotic Lactobacillus Zhang combined with routine treatment for gout hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion in this study only if they meet all of the following criteria

1. 18-70 years old, gender unlimited ；
2. Previous history of gout ；
3. According to the criteria of gout classification and diagnosis of EULAR / ACR in 2015；
4. fasting serum uric acid ≥ 480 μ mol / L (8mg / dl)

Exclusion Criteria:

If the subjects meet any of the following criteria, they will not be selected ：

1. Gout in the past two weeks ；
2. Secondary hyperuricemia ；
3. Patients with abnormal liver and kidney function (ALT, AST are 1.5 times higher than the normal value, Cr is 1.5 times higher than the upper limit of the normal value；
4. WBC < 4.0 × 109 / L, PLT < 100 × 109 / L, HGB < 90g / L, or other hematological diseases ；
5. bad blood pressure control (BP>160mmHg/100 mmHg)
6. Type I diabetes or poorly controlled type II diabetes: fasting blood glucose ≥ 8.5mmol/l ；
7. Patients with active peptic ulcer ；
8. Patients with gastrointestinal cancer ；
9. Patients with previous intestinal diseases such as lactose intolerance, irritable bowel syndrome, inflammatory bowel disease and habitual diarrhea ；
10. Use of drugs that affect the metabolism or excretion of uric acid and cannot / cannot be stopped, including azathioprine, 6-mercaptopterin, thiazide diuretics, aspirin (more than 325mg / day) or other salicylates ；
11. Those who need continuous prednisone treatment ；
12. Those who need antibiotic treatment for infectious diseases ；
13. Those with body mass index (BMI) greater than 30 ；
14. people with alcoholism ；
15. People with a history of allergy to Lactobacillus and its products or with high sensitive constitution ；
16. Researchers who have received other drugs within 3 months before screening ；
17. The people who are researchers thinks it is not suitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
serum uric acid level | 24 weeks
  The serum uric acid level was standard-reaching rate at the end of 24 weeks(Percentage of patients whose serum uric acid level has decreased to less than 360umol / L )

SECONDARY OUTCOMES:
serum uric acid level at the 4、8、12、24 weeks | 4、8、12、24 weeks
  the serum uric acid level and the percentage of patients with < 360umol / L at the end of 4, 8, 12 and 24 weeks after treatment
serum uric acid decreased from baseline | 4、8、12、24 weeks
  At the end of 4, 8, 12 and 24 weeks after treatment, the serum uric acid level decreased from baseline
Acute attack of gout | 24 week
  Number of acute gout attacks during 24 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Medical College Affiliated Hospital, Hohhot, Inner Mongolia, China